CLINICAL TRIAL: NCT00947492
Title: Monitoring EBV Load in Rheumatoid Arthritis Patients Treated With New Immunosuppressive Drugs ; Orencia* (Abatacept) and RoActemra* (Tocilizumab).
Brief Title: Monitoring Epstein-Barr Virus (EBV) Load in Rheumatoid Arthritis Patients Treated With New Immunosuppressive Drugs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2009-07; 2009-A00247-50
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis patients; treated with new immunosuppressive drugs : Orencia* (abatacept) and RoActemra* (tocilizumab).
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Venous blood sample — Venous blood sample twice a year during 3 years

SUMMARY:
PBMNC DNA is considered a limit above which patients will develop EBV associated post transplant lymphoproliferative disorder.

we showed that methotrexate tended to decrease EBV load over time, but this did not reach significance and that TNFa inhibitors did not significantly modify EBV load over time.

Our objective is to monitor Epstein Barr Virus load over time in patients with Rheumatoid arthritis under Orencia* (abatacept) or RoActemra* (tocilizumab), to detect possible immunosuppression associated EBV dysregulation, as seen in post transplant lymphoproliferative disease.

DETAILED DESCRIPTION:
Current treatment of RA routinely includes potentially immunosuppressive medications like methotrexate and TNFa inhibitors. New immunosuppressive drugs are at disposal, Orencia* (abatacept) which is a T cell co-stimulation modulator (CTLA4Ig) and RoActemra* (tocilizumab), an antibody against IL6 receptor. In solid organ transplant recipients under immunosuppressants, emergence of lymphoma can be predicted by monitoring EBV load in peripheral blood mononuclear cells (PBMNCs). EBV load above 1000 copies per 500 ng PBMNC DNA is considered a limit above which patients will develop EBV associated post transplant lymphoproliferative disorder, a condition characterized by polyclonal EBV positive B lymphocyte proliferation which can evolve into EBV positive B cell lymphoma .

In a first study, we showed that Rheumatoid arthritis patients have 10 fold systemic EBV overload, very similar to that observed in healthy organ transplant recipients. More recently, we showed that methotrexate tended to decrease EBV load over time, but this did not reach significance and that TNFa inhibitors did not significantly modify EBV load over time.

Our objective is to monitor Epstein Barr Virus load over time in patients with Rheumatoid arthritis under Orencia* (abatacept) or RoActemra* (tocilizumab), to detect possible immunosuppression associated EBV dysregulation, as seen in post transplant lymphoproliferative disease.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis patients
* treated with new immunosuppressive drugs : Orencia* (abatacept) and RoActemra* (tocilizumab)
* Disease longer than one year

Exclusion Criteria:

* Rheumatoid arthritis patients treated with ciclosporin in two years preceding the study
* Transplanted patients
* Disease shorter than one year
* Histories of lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-06; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
to monitor Epstein Barr Virus load over time in patients with Rheumatoid arthritis under Orencia* (abatacept) or RoActemra* (tocilizumab) | 3 years

SECONDARY OUTCOMES:
to detect possible immunosuppression associated EBV dysregulation, as seen in post transplant lymphoproliferative disease | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Balandraud, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique-Hopitaux de Marseille, Marseille, France